CLINICAL TRIAL: NCT04438694
Title: Assessment of the Effect of Convalescent Plasma Therapy in Patients With Life-threatening COVID19 Infection
Acronym: CP IN COVID19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen El Desouky, PROFESSOR OF CLINICAL PATHOLOGY, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N39-2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: COVID19
Keywords: DONOR; RECIPIENT; CONVALESCENT PLASMA
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-institution, single-arm, study using a historical control group for comparison. Open label, 2 arms: SOC and SOC+CP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STANDARD OF COARE (Active Comparator): Receiving SOC
  Interventions: Drug: Standard of Care
- STANDARD CP DOSE Adm (Two infusions) (Experimental): Two infusions 48 hours apart
  Interventions: Biological: Convalescent Plasma; Drug: Standard of Care

INTERVENTIONS:
Biological: Convalescent Plasma — Convalescent Plasma
  Arms: STANDARD CP DOSE Adm (Two infusions)
Drug: Standard of Care — Standard of Care drugs administered as per Cairo University ICU protocol

SUMMARY:
* This clinical trial proposal is based on the FDA protocol for emergency use of convalescent plasma for treatment of COVID-19 cases, and on the WHO guidelines for use of convalescent plasma in other infectious diseases.
* This Clinical trial is to be applied in Cairo University quarantine hospital. The collection, testing and storage of convalescent plasma will be done inside CUH main blood bank.

The concept of this clinical trial is built on the collection of convalescent plasma from individuals who had recovered from documented infection with SARS-CoV-2, to be used for patients with- or at high risk of progression to- severe/life-threatening clinical conditions due to SARS-CoV-2 infection.

An informed consent is required to join this clinical trial; patients will be transfused with one or two units of ABO compatible convalescent plasma. Those patients will be followed up and the clinical and laboratory data will be compiled, including adverse events related to the administration of convalescent plasma (CP).

Other data to be collected retrospectively will include patient demographics, acute care facility resource utilization (total length of stay, days in ICU, days intubated, and survival till discharge from an acute care facility).

DETAILED DESCRIPTION:
This study will be done inside Cairo university hospitals, it will involve a number of CP donors who were recovered from COVID-19 infection and were treated at Cairo University isolation hospital. The CP donation process will take place at CUH blood bank ,the number of the donors will be determined at the end of the study as it will vary according to the donation process .

The study will also include sixty seven /life threatening COVID-19 patients admitted to Cairo University isolation hospital.

ELIGIBILITY:
Inclusion Criteria:

* Must have laboratory confirmed COVID-19 and admitted to Cairo University isolation hospital.
* Admitted to acute care facility.
* Must have severe or immediately life-threatening COVID-19:

Severe disease is defined as:

* dyspnea,
* respiratory frequency ≥ 30/min,
* blood oxygen saturation ≤ 93%,
* partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300, and/or
* lung infiltrates > 50% within 24 to 48 hours (CT finding)

Life-threatening disease is defined as:

* respiratory failure,
* septic shock, and/or
* multiple organ dysfunction or failure

Exclusion Criteria:

* Pregnancy
* Autoimmune disorder
* Participated in a CP trial in the past 6 months

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization/Recovery status | 2-3 weeks
  Decrease of hospital days of safety until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No